CLINICAL TRIAL: NCT07291791
Title: Evaluation of the Neuromodulatory Effects of Transcranial Direct Current Stimulation on Pain in Knee Osteoarthritis Patients: A Double Blind Randomized Controlled Trial
Brief Title: tDCS for Pain Modulation in Knee Osteoarthritis
Acronym: KOA-tDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS121225
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Pain; Osteoarthritis; tDCS; Neuromodulation; Central Sensitization
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Two parallel arms: active tDCS and sham tDCS.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a participant- and assessor-blinded, sham-controlled clinical trial. All tDCS sessions will be delivered by a trained physiotherapist who is aware of group allocation, while both participants and the outcome assessor remain blinded. To maintain allocation concealment, the physiotherapist recorded each participant's assignment using coded geometric symbols, the meaning of which remained confidential until completion of data collection.
  Active and sham tDCS will be applied using identical electrode placements and device settings. In the sham condition, the current will be delivered for approximately 30 seconds and then gradually ramped down to zero to reproduce the initial tingling sensation of active stimulation, ensuring effective participant blinding. After all data are collected, group identities will be unmasked for statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants in this arm (active tDCS group) will receive active anodal transcranial direct current stimulation (tDCS) applied over the primary motor cortex (M1). Stimulation will be delivered at 2 mA for 20 minutes per session, for a total of 15 sessions (five sessions per week for three consecutive weeks). Electrode placement follows standardized M1 montage protocols.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants in this arm (sham tDCS group) will receive sham tDCS using identical electrode placement and device settings as the active tDCS arm. The current will be applied for approximately 30 seconds and then gradually ramped down to zero to mimic the initial tingling sensation of active stimulation while delivering no effective stimulation. A total of 15 sessions will be administered over three weeks.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Transcranial Direct Current Stimulation (tDCS) is a non-invasive neuromodulation technique that applies low-intensity direct current to modulate cortical excitability. In this trial, stimulation is delivered over the primary motor cortex (M1) using saline-soaked sponge electrodes. For the active arm, anodal tDCS is applied at 2 mA for 20 minutes per session, for 15 sessions over three weeks. For the sham arm, the same electrode placement and device settings are used, but the current is ramped down after approximately 30 seconds to mimic the sensation of active stimulation without producing neuromodulatory effects.
  Other Names: tDCS

SUMMARY:
Knee osteoarthritis (KOA) is a common condition that causes long-lasting knee pain and difficulty with daily activities. Many patients have pain that is stronger than expected from joint changes because the nervous system becomes more sensitive to pain. Transcranial direct current stimulation (tDCS) is a non-invasive technique that uses a small electrical current applied to the scalp to help reduce pain sensitivity.

This study will test whether active tDCS over the primary motor cortex can reduce pain and improve function in people with knee osteoarthritis. A total of 102 participants will be randomly assigned to receive either active tDCS or sham (placebo) stimulation. All participants will receive 15 sessions over three weeks. We will measure pain intensity, pain sensitivity, physical function, depression, cognition, and quality of life before the treatment, after the 3-week treatment program, and again at the 1-month follow-up.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a major cause of chronic pain, disability, and reduced quality of life. In many patients, the severity of pain exceeds structural joint damage due to peripheral and central sensitization, including impaired conditioned pain modulation (CPM). Such dysfunction in descending inhibitory pathways contributes to pain amplification and poor response to standard treatments. Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulatory technique capable of modulating cortical excitability, enhancing descending inhibition, and potentially restoring altered pain processing mechanisms.

This randomized, assessor- and participant-blinded, sham-controlled clinical trial will investigate the neuromodulatory effects of anodal primary motor cortex (M1) tDCS in patients with KOA exhibiting impaired CPM. A total of 102 participants who meet eligibility criteria will be randomly assigned (1:1) to receive either active anodal M1-tDCS (2 mA, 20 minutes per session) or sham stimulation, using identical electrode placement and brief initial stimulation to maintain blinding. Both groups will receive 15 sessions administered over three consecutive weeks.

Assessments will be conducted at baseline, immediately after the intervention, and at 1-month follow-up. Primary outcomes include changes in pain intensity measured by the Visual Analogue Scale (VAS) and Brief Pain Inventory (BPI). Secondary outcomes include peripheral and central sensitization measures-Pressure Pain Threshold (PPT), Conditioned Pain Modulation (CPM), Central Sensitization Inventory (CSI), and PainDETECT-as well as functional outcomes assessed using the WOMAC index, Timed Up and Go (TUG) test, and One-Leg Stance. Additional outcomes include depressive symptoms (Beck Depression Inventory, BDI), cognitive function (Mini-Mental State Examination, MMSE), and health-related quality of life (SF-12).

This study aims to provide a comprehensive evaluation of the analgesic and neuromodulatory effects of tDCS in KOA, and to clarify its impact on pain modulation, pain sensitization, physical function, depression, cognition, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis (KOA) according to the American College of Rheumatology (ACR) clinical criteria.
* Adults of both sexes aged 35 years or older.
* Clinical knee pain persisting for at least 3 months.
* Average knee pain intensity ≥ 4/10 on the Numerical Rating Scale (NRS; 0-10) during the previous 24 hours, with one dominant affected knee.
* Central sensitization phenotype: impaired conditioned pain modulation (CPM), defined as no change or a reduction in pressure pain threshold (PPT) after the conditioning stimulus, corresponding to a PPT ratio ≥ 1 (pre-to-post stimulus).
* Prior pharmacological pain management with NSAIDs and/or SNRIs discontinued due to adverse effects, intolerance, or contraindications, and able to complete the required washout period (2 weeks for NSAIDs and 4 weeks for SNRIs) before baseline assessment.
* Able and willing to provide written informed consent and comply with study procedures.

Exclusion Criteria:

Participants will be excluded if they have any condition that could affect cortical excitability, confound outcome measures, or interfere with tDCS safety, including:

* Other chronic pain conditions associated with central sensitization (e.g., fibromyalgia).
* Inflammatory arthropathies (e.g., rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus).
* Neuropathic pain syndromes (e.g., lumbar or cervical radiculopathy).
* Any clinically significant or unstable systemic disease (cardiovascular, hepatic, renal, or metabolic disorders).
* Pregnancy or active malignancy.
* Neurological or psychiatric disorders including epilepsy, history of syncope, traumatic brain injury with residual deficit, or major depressive disorder.
* Current participation in physiotherapy, electrotherapy, or exercise rehabilitation programs.
* Metallic implants or implanted electrical devices (e.g., pacemakers, cochlear implants, deep brain stimulators).
* Cognitive impairment interfering with understanding instructions or providing informed consent.
* Dermatological contraindications at stimulation or testing sites (e.g., open wounds, infection, irritation).
* History of alcohol or substance abuse, or current use of centrally acting medications that alter cortical excitability (e.g., benzodiazepines).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS and BPI Scores) | Baseline, immediately after the 15-session intervention, and at 1-month follow-up.
  Pain intensity will be assessed using the Visual Analogue Scale (VAS) and the Brief Pain Inventory (BPI). The primary outcome is the change in VAS and BPI pain scores from baseline to immediately post-intervention and one-month follow-up.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold (PPT) | Baseline, immediately after completing the 15 treatment sessions, and at 1-month follow-up
  PPT will be assessed using a digital pressure algometer at two standardized locations on the affected side-the medial knee joint line and the ipsilateral lower leg-to evaluate peripheral sensitization, as well as at a remote site on the forearm to assess central sensitization. The primary outcome will be the change in mean PPT values across three time points: baseline, immediately post-intervention, and 1-month follow-up.
Change in Central Sensitization using Central Sensitization Inventory (CSI) Score | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Central sensitization symptoms will be assessed using the Central Sensitization Inventory (CSI). The outcome is the change in CSI total score (0-100) between baseline, post-intervention, and follow-up.
Change in Conditioned Pain Modulation (CPM) Efficiency | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  CPM efficiency will be evaluated using the submaximal-effort tourniquet test. Pressure pain threshold (PPT) will be measured immediately before and after the conditioning stimulus. CPM efficiency will be calculated as the ratio of pre-conditioning PPT to post-conditioning PPT. A pre-to-post stimulus PPT ratio greater than or equal to 1 (indicating no change or a reduction in PPT after conditioning) will be classified as impaired CPM, reflecting deficient descending inhibitory pain modulation. The outcome is the change in CPM efficiency across baseline, post-intervention, and 1-month follow-up.
Change in neuropathic-like pain features (PainDETECT Score) | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Neuropathic-like pain features will be assessed using the PainDETECT questionnaire. The outcome is the change in PainDETECT total score across baseline, post-intervention, and follow-up.
Change in physical function (WOMAC Score) | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Pain, stiffness, and physical function will be evaluated using the WOMAC questionnaire. Higher WOMAC scores indicate greater physical dysfunction. The outcome is the change in WOMAC total and subscale scores from baseline to post-intervention and follow-up.
Change in functional performance using Timed Up and Go (TUG) Performance and One-Leg Stance (OLS) Time. | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Functional performance will be assessed using the Timed Up and Go (TUG) test for functional mobility and the One-Leg Stance (OLS) test for balance. The outcome is defined as the change in TUG completion time and the change in maximum OLS stance duration (in seconds) across baseline, post-intervention, and 1-month follow-up.
Change in depressive symptoms using the Beck Depression Inventory (BDI) Score | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Depressive symptoms will be assessed using the Beck Depression Inventory (BDI). The outcome is the change in total BDI score between baseline, post-intervention, and follow-up.
Change in cognitive function using Mini-Mental State Examination (MMSE) Score | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Cognitive function will be evaluated using the Mini-Mental State Examination (MMSE). The outcome is the change in MMSE score across baseline, post-intervention, and 1-month follow-up.
Change in SF-12 Quality of Life Score | Baseline, immediately after the 15-session intervention, and at 1-month follow-up
  Health-related quality of life will be assessed using the SF-12 questionnaire. The outcome is the change in physical and mental component summary scores from baseline to post-intervention and 1-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan E. Elkaraly, M.B.B.Ch.2015; MSc (PMRR)2020, Principal Investigator — Suez Canal University, Faculty of Medicine; Aziza S. Omar, M.D., Study Chair — Suez Canal University, Faculty of Medicine; Ahmed F. Genedy, M.D., Study Chair — Faculty of Medicine, Armed Forces Military Academy; Samah I. Nasef, M.D., Study Chair — Suez Canal University, Faculty of Medicine; Maha E. Ibrahim, M.D., Study Chair — Suez Canal University, Faculty of Medicine
Locations (1):
- Suez Canal University Hospitals - Physical Medicine, Rheumatology and Rehabilitation Outpatient Clinics, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center academic doctoral research project, and the ethical approval obtained does not permit public sharing of patient-level data. All collected data are confidential and will be used solely for the purposes of this study in accordance with institutional and national data protection regulations.